CLINICAL TRIAL: NCT00237692
Title: Behavioral/Pharmacological Telemedicine Interventions for BP Control
Brief Title: Hypertension Intervention Nurse Telemedicine Study (HINTS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IIR 04-426
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension
Keywords: Telemedicine; Adherence; Tailored Nurse Intervention; Home Blood Pressure Monitoring; cardiovascular disease
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (No Intervention): Control group - a group of hypertensive patient who receive usual care
- Arm 2 (Experimental): Nurse Behavioral intervention with Home BP Telemonitoring Nurse-administered tailored behavior intervention
  Interventions: Behavioral: Nurse Behavioral intervention with Home BP Telemonitoring
- Arm 3 (Experimental): Nurse Medication Management with Home BP Telemonitoring -- Nurse administer medication management according to hypertension decision support system
  Interventions: Behavioral: Nurse Medication Management with Home BP Telemonitoring
- Arm 4 (Experimental): Nurse Combined intervention with Home BP Telemonitoring - Combination of the nurse administered tailored behavioral & medication management interventions
  Interventions: Behavioral: Nurse Combined intervention with Home BP Telemonitoring

INTERVENTIONS:
Behavioral: Nurse Behavioral intervention with Home BP Telemonitoring — Nurse-administered behavior intervention
  Arms: Arm 2
Behavioral: Nurse Medication Management with Home BP Telemonitoring — Nurse administer medication management according to hypertension decision support
  Arms: Arm 3
Behavioral: Nurse Combined intervention with Home BP Telemonitoring — Combination of the nurse administered tailored behavioral & medication management
  Arms: Arm 4

SUMMARY:
There are 65 million Americans and over 8.5 million veterans who have been diagnosed with hypertension; yet only 31% of all hypertensive patients have their blood pressure (BP) under effective control (less than 140/90 mm/Hg). Uncontrolled hypertension greatly increases the risk of cerebral vascular accidents, coronary artery disease, myocardial infarction, renal failure, congestive heart failure, and mortality. Despite the damaging impact of hypertension and the availability of well-defined therapies and widely accepted target values for BP, interventions to improve BP control have had limited success.

DETAILED DESCRIPTION:
Detailed

Description Background:

There are 65 million Americans and over 8.5 million veterans who have been diagnosed with hypertension; yet only 31% of all hypertensive patients have their blood pressure (BP) under effective control (<140/90 mm/Hg). Uncontrolled hypertension greatly increases the risk of cerebral vascular accidents, coronary artery disease, myocardial infarction, renal failure, congestive heart failure, and mortality. Despite the damaging impact of hypertension and the availability of well-defined therapies and widely accepted target values for BP, interventions to improve BP control have had limited success.

Objectives:

The study is one of the first to compare three interventions designed to improve BP control: a behavioral educational intervention, an evidence-based medication management intervention, and combined intervention for patients with poor BP control defined by home BP monitoring. The primary hypotheses are: 1) Patients who receive only the behavioral intervention will show improved rates of BP control as compared to the control group over 18 months of follow-up; 2) Patients who receive only the hypertension medication management intervention will show improved rates of BP control as compared to the control group over 18 months of follow-up; and, 3) Patients who receive the combined intervention will show higher rates of BP control as compared to all other patients over the 18 months of follow-up.

Methods:

A three-year randomized controlled trial among veterans with poor BP control testing three interventions in three VA primary care clinics is proposed to improve BP control. We will test these interventions using home BP monitoring in a four group design administered via the telephone: 1) control group - a group of hypertensive patients who receive usual care; 2) Nurse-administered tailored behavioral intervention previously tested (HSR&D grant IIR 20-034); 3) Nurse-administered medication management according to a hypertension decision support system that uses the VA's Computerized Medical Record System (VA HSR&D grant CPI 99275); 4) combination of the tailored behavioral and medication management interventions.

A random sample of hypertensive patients with poor BP control at baseline were consented and randomly allocated to one of four arms. The interventions will activate only when home BP monitoring indicates inadequate BP control. Patients assigned to the behavioral intervention will receive a tailored self-management intervention to promote adherence with medication, information on the risks of hypertension and health behaviors at periodic telephone contacts. Patients will receive feedback about their recent BP values, continuous patient education, and will be monitored and supported to enhance treatment adherence. Patients randomized to the medication management arm will have their hypertension regimen changed by a nurse using a hypertension decision support system developed and validated in the VA. Medication recommendations generated are based on JNC 7 and the VA's hypertension treatment guidelines and are also individualized to patients' comorbid illnesses, laboratory values, and other elements of patients' clinical status. Medication management will be based on home BP monitoring and delivered by telephone. The nurse is part of an extended primary care team and communicates changes to the patients' primary care providers via a study physician.

The primary outcome will be a dichotomous measure representing whether or not the patient's BP is in control: >140/90 mm/Hg (non-diabetic) and >130/80 mm/Hg (diabetics). Measures will be made at six-month intervals over 18 months (4 total measurements). We will model the outcome measures and evaluate the interventions using a mixed effects model for dichotomous outcomes.

Status:

Primary study enrollment began May 5, 2006 and was completed November 2007. We randomized 591 participants in the study. Baseline recruitment was completed in November 2007. Participants' completed the six month follow-up interviews in June 2008 and 12 month follow-up in December 2008. 18 month follow-up was completed June 2009.

Study was granted an extension to complete two goals: 1) investigate the sustainability of BP control after completion of intervention, and , 2) examine what aspects of the intervention worked or did not work using qualitative interviews.

Background/Rationale:

Despite the impact of hypertension and the availability of well-defined therapies and widely accepted target values for blood pressure (BP), interventions to improve BP control have had limited success.

Objectives:

The study is one of the first to compare three interventions designed to improve BP control: a behavioral educational intervention, an evidence-based medication management intervention, and combined intervention for patients with poor BP control defined by home BP monitoring. We received an 11 month extension to evaluate 3 key components of the study (sustainability of BP effects, qualitative evaluation of the intervention, evaluation of the supporting materials used to ensure literacy levels and cultural sensitivity.)

Methods:

A 4-arm randomized trial with 18-month follow-up. Patents were selected from primary care clinics at the Durham VA Medical Center. Of the eligible patients, 591 individuals were randomized to either usual care or one of three telephone-based intervention groups. The intervention phone calls were triggered based on home BP values transmitted via telemonitoring devices. Patients were instructed to take their BP three times a week and transmit to study team. Behavioral management involved promoting health behaviors. Medication management involved adjustment of hypertension medications by a study physician and nurse based on hypertension treatment guidelines. The primary outcome was changes in BP control measured at six-month intervals over 18 months. For the sustainability extension of the study, in additional to collection of BP values, we will use qualitative analysis to examine the audio interviews.

Status:

Sustainability phase recruitment began May 1, 2010 and ended on Aug 15, 2010. Analyses are continuing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of uncontrolled hypertension,
* prescribed a medication to lower blood pressure,
* have a regular primary care physician at Durham VA Medical Center, and
* be a veteran. For Sustainability portion the patient must have participated in an intervention arm of primary study.

Exclusion Criteria:

* Hospitalized in past 3 months for stroke,
* heart attack,
* surgery for blocked arteries,
* diagnosed with metastatic cancer or treated with dialysis,
* have a diagnosis of dementia or a hearing impairment which prevents them from being able to hear/speak on the telephone, and
* creatinine serum lab which exceed 2.5.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 591 (Actual)
Dates: Start 2006-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hayden B. Bosworth, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Background] Bosworth HB, Olsen MK, McCant F, Harrelson M, Gentry P, Rose C, Goldstein MK, Hoffman BB, Powers B, Oddone EZ. Hypertension Intervention Nurse Telemedicine Study (HINTS): testing a multifactorial tailored behavioral/educational and a medication management intervention for blood pressure control. Am Heart J. 2007 Jun;153(6):918-24. doi: 10.1016/j.ahj.2007.03.004. PMID 17540191
- [Result] Crowley MJ, Grubber JM, Olsen MK, Bosworth HB. Factors associated with non-adherence to three hypertension self-management behaviors: preliminary data for a new instrument. J Gen Intern Med. 2013 Jan;28(1):99-106. doi: 10.1007/s11606-012-2195-1. Epub 2012 Aug 28. PMID 22926634
- [Result] Jackson GL, Oddone EZ, Olsen MK, Powers BJ, Grubber JM, McCant F, Bosworth HB. Racial differences in the effect of a telephone-delivered hypertension disease management program. J Gen Intern Med. 2012 Dec;27(12):1682-9. doi: 10.1007/s11606-012-2138-x. Epub 2012 Aug 3. PMID 22865016
- [Result] Wang V, Smith VA, Bosworth HB, Oddone EZ, Olsen MK, McCant F, Powers BJ, Van Houtven CH. Economic evaluation of telephone self-management interventions for blood pressure control. Am Heart J. 2012 Jun;163(6):980-6. doi: 10.1016/j.ahj.2012.03.016. Epub 2012 May 21. PMID 22709750
- [Result] Crowley MJ, Smith VA, Olsen MK, Danus S, Oddone EZ, Bosworth HB, Powers BJ. Treatment intensification in a hypertension telemanagement trial: clinical inertia or good clinical judgment? Hypertension. 2011 Oct;58(4):552-8. doi: 10.1161/HYPERTENSIONAHA.111.174367. Epub 2011 Aug 15. PMID 21844490
- [Result] Bosworth HB, Powers BJ, Olsen MK, McCant F, Grubber J, Smith V, Gentry PW, Rose C, Van Houtven C, Wang V, Goldstein MK, Oddone EZ. Home blood pressure management and improved blood pressure control: results from a randomized controlled trial. Arch Intern Med. 2011 Jul 11;171(13):1173-80. doi: 10.1001/archinternmed.2011.276. PMID 21747013
- [Result] Powers BJ, Olsen MK, Smith VA, Woolson RF, Bosworth HB, Oddone EZ. Measuring blood pressure for decision making and quality reporting: where and how many measures? Ann Intern Med. 2011 Jun 21;154(12):781-8, W-289-90. doi: 10.7326/0003-4819-154-12-201106210-00005. PMID 21690592
- [Result] Powers BJ, Danus S, Grubber JM, Olsen MK, Oddone EZ, Bosworth HB. The effectiveness of personalized coronary heart disease and stroke risk communication. Am Heart J. 2011 Apr;161(4):673-80. doi: 10.1016/j.ahj.2010.12.021. PMID 21473965
- [Result] Zullig LL, Melnyk SD, Goldstein K, Shaw RJ, Bosworth HB. The role of home blood pressure telemonitoring in managing hypertensive populations. Curr Hypertens Rep. 2013 Aug;15(4):346-55. doi: 10.1007/s11906-013-0351-6. PMID 23625207
- [Result] Bowen ME, Bosworth HB, Roumie CL. Blood pressure control in a hypertension telemedicine intervention: does distance to primary care matter? J Clin Hypertens (Greenwich). 2013 Oct;15(10):723-30. doi: 10.1111/jch.12172. Epub 2013 Jul 23. PMID 24088280
- [Result] Bosworth HB, Olsen MK, Dudley T, Orr M, Goldstein MK, Datta SK, McCant F, Gentry P, Simel DL, Oddone EZ. Patient education and provider decision support to control blood pressure in primary care: a cluster randomized trial. Am Heart J. 2009 Mar;157(3):450-6. doi: 10.1016/j.ahj.2008.11.003. Epub 2009 Jan 10. PMID 19249414
- [Result] McCant F, McKoy G, Grubber J, Olsen MK, Oddone E, Powers B, Bosworth HB. Feasibility of blood pressure telemonitoring in patients with poor blood pressure control. J Telemed Telecare. 2009;15(6):281-5. doi: 10.1258/jtt.2009.090202. PMID 19720764
- [Derived] Maciejewski ML, Bosworth HB, Olsen MK, Smith VA, Edelman D, Powers BJ, Kaufman MA, Oddone EZ, Jackson GL. Do the benefits of participation in a hypertension self-management trial persist after patients resume usual care? Circ Cardiovasc Qual Outcomes. 2014 Mar;7(2):269-75. doi: 10.1161/CIRCOUTCOMES.113.000309. Epub 2014 Mar 11. PMID 24619321

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1- Control: A group of hypertensive patients who receive usual care
- Arm 2 - Nurse Behavioral Int: Nurse Behavioral intervention with Home BP Telemonitoring: Nurse-administered behavior intervention
- Arm 3 - Nurse Med Managment Int: Nurse Medication Management with Home BP Telemonitoring: Nurse administer medication management according to hypertension decision support
- Arm 4 - Combined Behavioral and Med Mgmt Int: Nurse Combined intervention with Home BP Telemonitoring: Combination of the nurse administered tailored behavioral & medication management
Period: Overall Study
Arm/Group | Arm 1- Control | Arm 2 - Nurse Behavioral Int | Arm 3 - Nurse Med Managment Int | Arm 4 - Combined Behavioral and Med Mgmt Int
Started | 147 | 148 | 149 | 147
6 Month f/u | 132 | 134 | 135 | 134
12 Month f/u | 137 | 127 | 132 | 127
18 Month f/u | 124 | 131 | 126 | 122
Completed | 129 | 134 | 127 | 128
Not Completed | 18 | 14 | 22 | 19
Not completed — Lost to Follow-up | 9 | 3 | 5 | 3
Not completed — Death | 1 | 2 | 2 | 3
Not completed — Excluded - did not meet criteria | 4 | 3 | 5 | 9
Not completed — Withdrawal by Subject | 4 | 6 | 10 | 4

BASELINE CHARACTERISTICS:
Population: All data except blood pressure, age, gender were patient-reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1- Control | Arm 2 - Nurse Behavioral Int | Arm 3 - Nurse Med Managment Int | Arm 4 - Combined Behavioral and Med Mgmt Int | Total
Number analyzed (Participants) | 147 | 148 | 149 | 147 | 591
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10) | 63 (11) | 64 (10) | 63 (11) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 10 | 21 | 49
  Male | 141 | 136 | 139 | 126 | 542
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 74 | 78 | 73 | 64 | 289
  African American | 71 | 66 | 72 | 76 | 285
  Other | 2 | 4 | 4 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 147 | 148 | 149 | 147 | 591

OUTCOME MEASURES:

1. Primary Outcome: Estimated Percentage of Participants in Blood Pressure Control at Baseline
Description: When patients had multiple blood pressure readings during their baseline visit, means of their systolic and diastolic readings were used as the baseline blood pressure values; Using Joint National Committee 7 Report (JNC7) blood pressure guidelines for BP control: <140/90mmHg for non-diabetic patients and < 130/80mmHg for diabetic patients
Time Frame: Baseline
Measure: Number; unit: % of particpants w/ controlled BP
Groups:
- Arm 3 - Nurse Med Management Int: Nurse Medication Management with Home BP Telemonitoring: Nurse administer medication management according to hypertension decision support
- Arm 4 - Combined Behaviorial and Med Mgmt Int: Nurse Combined intervention with Home BP Telemonitoring: Combination of the nurse administered tailored behavioral & medication management
Arm/Group | Arm 1- Control | Arm 2 - Nurse Behavioral Int | Arm 3 - Nurse Med Management Int | Arm 4 - Combined Behaviorial and Med Mgmt Int
Number analyzed (Participants) | 147 | 148 | 149 | 147
% of particpants w/ controlled BP | 61 | 59 | 53 | 64
Statistical Analysis 1: Comparison: Arm 1- Control; Estimated % of participants with controlled Systolic BP at Baseline; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 59.8, 95% CI 2-sided [55.7 to 63.9] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 2: Comparison: Arm 2 - Nurse Behavioral Int; Estimated % of participants with controlled Systolic BP at Baseline; Test type: Superiority or Other; Est. % of patients with controled SBP = 59.8, 95% CI 2-sided [55.7 to 64.0] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 3: Comparison: Arm 3 - Nurse Med Management Int; Estimated % of participants with controlled BP at Baseline; Test type: Superiority or Other; Est. % of patinets with controlled SBP = 59.8, 95% CI 2-sided [55.6 to 63.9] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 4: Comparison: Arm 4 - Combined Behaviorial and Med Mgmt Int; Estimated % of participants with controlled Systolic BP at Baseline; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 59.8, 95% CI 2-sided [55.6 to 63.9] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics

2. Primary Outcome: Estimated Percentage of Participants in Blood Pressure Control at 6 Months
Description: When patients had multiple blood pressure readings during their 6 month visit, means of their systolic and diastolic readings were used as the 6 month blood pressure values; Using Joint National Committee 7 Report (JNC7) blood pressure guidelines for BP control: <140/90mmHg for non-diabetic patients and < 130/80mmHg for diabetic patients
Time Frame: 6month
Measure: Number; unit: % of particpants with controlled SBP
Arm/Group | Arm 1- Control | Arm 2 - Nurse Behavioral Int | Arm 3 - Nurse Med Management Int | Arm 4 - Combined Behaviorial and Med Mgmt Int
Number analyzed (Participants) | 132 | 134 | 135 | 134
% of particpants with controlled SBP | 58 | 61 | 65 | 64
Statistical Analysis 1: Comparison: Arm 1- Control; Estimated % of participants with controlled Systolic BP at 6 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 58.0, 95% CI 2-sided [49.3 to 66.7] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 2: Comparison: Arm 2 - Nurse Behavioral Int; Estimated % of participants with controlled systolic BP at 6 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 60.9, 95% CI 2-sided [52.5 to 69.3] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 3: Comparison: Arm 3 - Nurse Med Management Int; Estimated % of participants with controlled systolic BP at 6 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 65.0, 95% CI 2-sided [56.9 to 73.1] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 4: Comparison: Arm 4 - Combined Behaviorial and Med Mgmt Int; Estimated % of participants with controlled systolic BP at 6 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 63.8, 95% CI 2-sided [55.6 to 72.0] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 5: Comparison: Arm 1- Control vs Arm 2 - Nurse Behavioral Int; Estimated Difference in Percentage of Patients with Controlled Systolic Blood pressure between Intervention Arm 2 - Nurse Behavioral and Arm 1 - Control at 6months; Test type: Superiority or Other; % diff = 2.9, 95% CI 2-sided [-9.0 to 14.9] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 6: Comparison: Arm 1- Control vs Arm 3 - Nurse Med Management Int; Estimated Difference in Percentage of Patients with Controlled Systolic Blood pressure between Intervention Arm 2 - Nurse Med Management and Arm 1 - Control at 6months; Test type: Superiority or Other; % Diff = 6.9, 95% CI 2-sided [-4.7 to 18.7] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 7: Comparison: Arm 1- Control vs Arm 4 - Combined Behaviorial and Med Mgmt Int; Estimated Difference in Percentage of Patients with Controlled Systolic Blood pressure between Intervention Arm 2 - Combined Behavioral & Med Mgmt and Arm 1 - Control at 6months; Test type: Superiority or Other; % Diff = 5.7, 95% CI 2-sided [-6.0 to 17.6]

3. Primary Outcome: Estimated Percentage of Participants in Blood Pressure Control at 12 Months
Description: When patients had multiple blood pressure readings during their 12 month visit, means of their systolic and diastolic readings were used as the 12 month blood pressure values; Using Joint National Committee 7 Report (JNC7) blood pressure guidelines for BP control: <140/90mmHg for non-diabetic patients and < 130/80mmHg for diabetic patients
Time Frame: 12 month
Measure: Number; unit: % of particpants with controlled SBP
Arm/Group | Arm 1- Control | Arm 2 - Nurse Behavioral Int | Arm 3 - Nurse Med Management Int | Arm 4 - Combined Behaviorial and Med Mgmt Int
Number analyzed (Participants) | 137 | 127 | 132 | 127
% of particpants with controlled SBP | 60 | 73 | 73 | 69
Statistical Analysis 1: Comparison: Arm 1- Control; Estimated % of participants with controlled systolic BP at 12 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 59.9, 95% CI 2-sided [51.4 to 68.3] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 2: Comparison: Arm 2 - Nurse Behavioral Int; Estimated % of participants with controlled systolic BP at 12 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 73.1, 95% CI 2-sided [65.6 to 80.7] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 3: Comparison: Arm 3 - Nurse Med Management Int; Estimated % of participants with controlled systolic BP at 12 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 73.4, 95% CI 2-sided [66.1 to 80.7] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 4: Comparison: Arm 4 - Combined Behaviorial and Med Mgmt Int; Estimated % of participants with controlled Systolic BP at 12 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 68.6, 95% CI 2-sided [60.5 to 76.6] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 5: Comparison: Arm 1- Control vs Arm 2 - Nurse Behavioral Int; Estimated Difference in Percentage of Patients with Controlled Systolic Blood pressure between Intervention Arm 2 - Nurse Behavioral and Arm 1 - Control at 12 months; Test type: Superiority or Other; % Diff = 13.2, 95% CI 2-sided [2.0 to 24.4]
Statistical Analysis 6: Comparison: Arm 1- Control vs Arm 3 - Nurse Med Management Int; Estimated Difference in Percentage of Patients with Controlled Systolic Blood pressure between Intervention Arm 3 - Nurse Med Management and Arm 1 - Control at 12 months; Test type: Superiority or Other; % Diff = 13.5, 95% CI 2-sided [2.4 to 24.6]
Statistical Analysis 7: Comparison: Arm 1- Control vs Arm 4 - Combined Behaviorial and Med Mgmt Int; Estimated Difference in Percentage of Patients with Controlled Systolic Blood pressure between Intervention Arm 4 - Combined Behavioral & Med Mgmt and Arm 1 - Control at 12 months; Test type: Superiority or Other; % diff = 8.6, 95% CI 2-sided [-2.9 to 20.2]

4. Primary Outcome: Estimated Percentage of Participants in Blood Pressure Control at 18 Months
Description: When patients had multiple blood pressure readings during their 18 month visit, means of their systolic and diastolic readings were used as the 18 month blood pressure values; Using Joint National Committee 7 Report (JNC7) blood pressure guidelines for BP control: <140/90mmHg for non-diabetic patients and < 130/80mmHg for diabetic patients
Time Frame: 18 month
Measure: Number; unit: % of particpants with controlled SBP
Arm/Group | Arm 1- Control | Arm 2 - Nurse Behavioral Int | Arm 3 - Nurse Med Management Int | Arm 4 - Combined Behaviorial and Med Mgmt Int
Number analyzed (Participants) | 124 | 131 | 126 | 122
% of particpants with controlled SBP | 62 | 59 | 64 | 72
Statistical Analysis 1: Comparison: Arm 1- Control; Estimated % of participants with controlled Systolic BP at 18 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 61.8, 95% CI 2-sided [53.0 to 70.6] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 2: Comparison: Arm 2 - Nurse Behavioral Int; Estimated % of participants with controlled BP at 18 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 59.4, 95% CI 2-sided [50.8 to 67.9] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 3: Comparison: Arm 3 - Nurse Med Management Int; Estimated % of participants with controlled systolic BP at 18 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 63.5, 95% CI 2-sided [55.1 to 72.0] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 4: Comparison: Arm 4 - Combined Behaviorial and Med Mgmt Int; Estimated % of participants with controlled systolic BP at 18 months; Test type: Superiority or Other; Est. % of Patients with controlled SBP = 71.6, 95% CI 2-sided [63.7 to 79.5] — Joint National Committee 7 blood pressure control: < 140/90 mmHg for non-diabetics; <130/80 mmHg for diabetics
Statistical Analysis 5: Comparison: Arm 1- Control vs Arm 2 - Nurse Behavioral Int; Estimated Difference in Percentage of Patients with Controlled Systolic Blood pressure between Intervention Arm 2 - Nurse Behavioral and Arm 1 - Control at 18 months; Test type: Superiority or Other; % Diff = -2.4, 95% CI 2-sided [-14.6 to 9.7]
Statistical Analysis 6: Comparison: Arm 1- Control vs Arm 3 - Nurse Med Management Int; Estimated Difference in Percentage of Patients with Controlled Systolic Blood pressure between Intervention Arm 3 - Nurse Med Management and Arm 1 - Control at 18 months; Test type: Superiority or Other; % Diff = 1.7, 95% CI 2-sided [-10.3 to 13.8]
Statistical Analysis 7: Comparison: Arm 1- Control vs Arm 4 - Combined Behaviorial and Med Mgmt Int; Estimated Difference in Percentage of Patients with Controlled Systolic Blood pressure between Intervention Arm 4 - Combined Behavioral & Med Mgmt and Arm 1 - Control at 18 months; Test type: Superiority or Other; % Diff = 9.8, 95% CI 2-sided [-1.9 to 21.4]

5. Primary Outcome: Blood Pressure Averages Systolic & Diastolic
Description: Blood pressure measured at Baseline.
  BP control estimates are marginalized probabilities with corresponding 95% confidence intervals derived from a logistic mixed effects regression model.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1- Control | Arm 2 - Nurse Behavioral Int | Arm 3 - Nurse Med Management Int | Arm 4 - Combined Behaviorial and Med Mgmt Int
Number analyzed (Participants) | 147 | 148 | 149 | 147
mmHg
  Systolic BP | 128 (17) | 129 (19) | 132 (21) | 127 (21)
  Diastolic BP | 78 (14) | 77 (12) | 78 (14) | 77 (13)

6. Primary Outcome: Blood Pressure Averages Systolic & Diastolic
Description: Blood pressure measured at 12 month.
  BP control estimates are marginalized probabilities with corresponding 95% confidence intervals derived from a logistic mixed effects regression model.
Time Frame: 12-month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1- Control | Arm 2 - Nurse Behavioral Int | Arm 3 - Nurse Med Management Int | Arm 4 - Combined Behaviorial and Med Mgmt Int
Number analyzed (Participants) | 137 | 127 | 132 | 127
mmHg
  Systolic BP | 127.1 (1.5) | 125.0 (1.5) | 124.7 (1.5) | 122.8 (1.5)
  Diastolic BP | 75.6 (.9) | 74.9 (.9) | 74.6 (.9) | 75.6 (.9)
Statistical Analysis 1: Comparison: Arm 1- Control vs Arm 2 - Nurse Behavioral Int; Estimated differences in systolic blood pressure at 12months between Arm 1 - Control and Arm 2 - Nurse Behavioral; Test type: Superiority or Other; Est. % Diff in Patient w/Controlled SBP = 2.0, 95% CI 2-sided [-3.1 to 7.1] — Systolic blood pressure estimates are based on the longitudinal data model with an unstructured covariance matrix. Negative differences reflect improvement compared to usual care, and positive differences reflect worsening compared to usual care
Statistical Analysis 2: Comparison: Arm 1- Control vs Arm 2 - Nurse Behavioral Int; Estimated differences in diastolic blood pressure at 12months between Arm 1 - Control and Arm 2 - Nurse Behavioral; Test type: Superiority or Other; Est. Dif in Patient w/Controlled DBP = .5, 95% CI 2-sided [-2.7 to 3.8] — Diastolic blood pressure estimates are based on the longitudinal data model with an unstructured covariance matrix. Negative differences reflect improvement compared to usual care, and positive differences reflect worsening compared to usual care
Statistical Analysis 3: Comparison: Arm 1- Control vs Arm 3 - Nurse Med Management Int; Estimated differences in systolic blood pressure at 12months between Arm 1 - Control and Arm 3 - Nurse Med Management; Test type: Superiority or Other; Est. % Diff in Patient w/Controlled SBP = 0.4, 95% CI 2-sided [-4.8 to 5.5] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Arm 1- Control vs Arm 3 - Nurse Med Management Int; Estimated differences in diastolic blood pressure at 12months between Arm 1 - Control and Arm 3 - Nuse Med Management; Test type: Superiority or Other; Est. % Diff in Patient w/Controlled DBP = 0.7, 95% CI 2-sided [-2.6 to 4.0] — [estimate comment as in outcome 6, analysis 2]
Statistical Analysis 5: Comparison: Arm 1- Control vs Arm 4 - Combined Behaviorial and Med Mgmt Int; Estimated differences in systolic blood pressure at 12months between Arm 1 - Control and Arm 4 - Combined Behaviorial and Med Management; Test type: Superiority or Other; Est. % Diff in Patient w/Controlled SBP = 1.6, 95% CI 2-sided [-3.3 to 6.6] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Arm 1- Control vs Arm 4 - Combined Behaviorial and Med Mgmt Int; Estimated differences in diastolic blood pressure at 12months between Arm 1 - Control and Arm 4 - Combined Behaviorial and Med Management; Test type: Superiority or Other; Est. % Diff in Patient w/Controlled DBP = 3.4, 95% CI 2-sided [0.3 to 6.6] — [estimate comment as in outcome 6, analysis 2]

ADVERSE EVENTS:
Time Frame: Overall length of study
Arm/Group | Arm 1- Control | Arm 2 - Nurse Behavioral Int | Arm 3 - Nurse Med Managment Int | Arm 4 - Combined Behavioral and Med Mgmt Int
Serious Adverse Events (participants affected / at risk) | 43/147 | 71/148 | 68/149 | 60/147
Other Adverse Events (participants affected / at risk) | 0/147 | 0/148 | 0/149 | 0/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1- Control (N=147) | Arm 2 - Nurse Behavioral Int (N=148) | Arm 3 - Nurse Med Managment Int (N=149) | Arm 4 - Combined Behavioral and Med Mgmt Int (N=147)
w/recurrent nosebleed (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer Tx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Circulatory (Blood and lymphatic system disorders) | 3 (4) | 6 (6) | 6 (7) | 1 (1)
Coronary (Cardiac disorders) | 9 (9) | 18 (21) | 20 (26) | 11 (18)
Dermatologic (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (7) | 3 (3) | 3 (3)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1)
Endocrine (Endocrine disorders) | 4 (5) | 11 (18) | 7 (15) | 7 (7)
Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastro-Intestinal (Gastrointestinal disorders) | 3 (3) | 15 (30) | 11 (17) | 6 (6)
General - ER visits (General disorders) | 5 (5) | 2 (2) | 7 (8) | 3 (3)
General - Med-Refill (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
General - Med Side Effect (General disorders) | 3 (3) | 1 (1) | 4 (4) | 5 (5)
Infections (Infections and infestations) | 9 (11) | 8 (9) | 12 (12) | 9 (17)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Neurologic (Nervous system disorders) | 1 (1) | 8 (9) | 10 (11) | 5 (5)
Optometry (Eye disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Orthopedic Issues (Musculoskeletal and connective tissue disorders) | 11 (17) | 15 (22) | 18 (26) | 21 (30)
Psychological (Psychiatric disorders) | 2 (3) | 5 (5) | 3 (4) | 3 (5)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 17 (21) | 13 (20) | 9 (10)
Pulmonary-Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urology (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Vascular (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Coronary - Death (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Coronary Safety Protocol (Cardiac disorders) | 1 (1) | 1 (1) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No